CLINICAL TRIAL: NCT05792826
Title: Efficacy and Safety of BSZY Cream for Atopic Facial Dermatitis: a Randomized, Double-blind, Controlled Trial.
Brief Title: Clinical Study of BSZY Cream Intervention to Relieve Atopic Facial Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-024
Record Dates: First submitted 2023-02-08; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis of Face (Diagnosis)
Keywords: atopic facial dermatitis.
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BSZY Cream group (Experimental): receiving BSZY Cream twice a day,in the morning and evening, for a period of four weeks.
  Interventions: Other: BSZY Cream
- emulsion matrix group (Placebo Comparator): receiving the emulsion base twice a day, in the morning and evening, for a period of four weeks.
  Interventions: Other: emulsion matrix

INTERVENTIONS:
Other: BSZY Cream — The patients receive BSZY Cream twice a day, in the morning and evening, for a period of four weeks.The patients can continue using their usual sunscreen and cleansing products, and their skin care steps should follow their daily habits. It is not recommended to add or replace any previously unused skin care products during the testing period.
  Arms: BSZY Cream group
Other: emulsion matrix — The patients receive emusion matrix twice a day, in the morning and evening, for a period of four weeks.The patients can continue using their usual sunscreen and cleansing products, and their skin care steps should follow their daily habits. It is not recommended to add or replace any previously unused skin care products during the testing period.
  Arms: emulsion matrix group

SUMMARY:
This randomized double-blind controlled trial will be conducted in conducted in the Department of Dermatology at the Yueyang Hospital of Integrated Traditional Chinese and Western Medicine in China.An estimated 130 participants will be recruited and randomly assigned to receive BSZY Cream or emulsion matrix group in a l:l ratio using SPSS 25.0 software.Application is twice a day, morning and evening, for four weeks.The primary outcome will be the SCORAD scale.The secondary outcomes included clinical dermatologist assessment forms, patient self-assessment questionnaires, and safety indicators.The adverse events will be recorded for safety evaluation. All data in the study will be analyzed using the SPSS 25.0 statistical software package.

DETAILED DESCRIPTION:
This randomized, double-blind, controlled trial will be conducted at Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine. Trials will begin following ethics approval and protocol registration. Patient recruitment began in April 2023 and is expected to conclude in June 2024. An estimated 130 participants will be enrolled and randomized 1:1 to receive BSZY Cream or emulsion base. In the process of developing standard protocols, the Standards for Reporting Interventions in Clinical Trials of Acupuncture and Moxibustion (STRICTA) and the SPIRIT Reporting Guidelines will be followed to clearly and transparently explain the treatment process involved.

Potential subjects were assessed for eligibility for inclusion and exclusion criteria. Eligible participants will voluntarily provide written informed consent prior to randomization.

This study will use a double-blind design. Both BSZY Cream and emulsion base were provided by the manufacturer, and were distributed by designated research nurses after registration, once every 2 weeks. Except for the first dispensing, the unused lotion was collected and counted each time after dispensing.

ELIGIBILITY:
Inclusion Criteria:

The general inclusion criteria for the study are as follows:

1. Meet the diagnostic criteria for patients with atopic dermatitis in the China Atopic Dermatitis Treatment Guidelines (2020 Edition);
2. Age ≥ 18 years old;
3. Able to cooperate with receiving topical cream treatment;
4. Voluntary participation in clinical trial studies and signing of informed consent (informed consent signed by the patient, legal guardian or person in charge of the medical situation via paper signature);
5. Willingness to replace the test product with a cream-based product currently in use. Not be recommended to use their own skin care products in that dosage form throughout the testing period;
6. Facial manifestations of atopic dermatitis.

Exclusion Criteria:

1. Previous allergies to ingredients such as skin care products, soaps, alcohol, fragrances or medications;
2. Insulin-dependent diabetic patients;
3. Received anti-cancer chemotherapy within the last 6 months;
4. Patients with immune deficiencies or autoimmune diseases;
5. Lactating or pregnant women;
6. Bilateral mastectomy and bilateral axillary lymph node dissection;
7. Subjects with observed facial wounds, abrasions, tattoos, or other conditions affecting the determination of test results;
8. Have participated in outdoor, travel and other high-intensity sun exposure activities that may cause skin damage in the month prior to the test;
9. Those who are also participating in another clinical test or have participated in a facial clinical test within the last three months;
10. Vitamin A, a hydroxy acid, salicylic acid, hydroquinone applied within the last 3 months, or prescription drugs (antibiotics, vitamin A, a hydroxy acid and steroids) within the last 6 months, oral contraceptives (if you have been taking the same type of contraceptive for the last 6 months, you can continue to take them);
11. Clinical dermatologists or professionals believe there are other medical reasons that could affect the test results;
12. SCORAD score >50 (atopic dermatitis SCORAD score: mild: 0~24, moderate: 25~50, severe: >50).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
SCORAD | At weeks 0 after the patient's admission
  The SCORAD score was calculated based on the types of lesions and body areas and was assessed separately for the head, neck, arms, legs, anterior trunk, back, and genitalia based on the area of skin involved and the severity of erythema, exudation, crusting, lichenification, and dryness. The scores report the severity of the patients' symptoms, with a total score ranging from 0 to 103, scores of 25 or lower indicating mild severity, scores of 26 to 50 indicating moderate severity, and scores of 51 to 103 indicating severe severity.. Patients were monitored for changes in SCROAD during treatment, observed for improvement in atopic dermatitis, and changes in points were calculated and compared before and after.
SCORAD | At weeks 2 after the patient's admission
  The SCORAD score was calculated based on the types of lesions and body areas and was assessed separately for the head, neck, arms, legs, anterior trunk, back, and genitalia based on the area of skin involved and the severity of erythema, exudation, crusting, lichenification, and dryness. The scores report the severity of the patients' symptoms, with a total score ranging from 0 to 103, scores of 25 or lower indicating mild severity, scores of 26 to 50 indicating moderate severity, and scores of 51 to 103 indicating severe severity.. Patients were monitored for changes in SCROAD during treatment, observed for improvement in atopic dermatitis, and changes in points were calculated and compared before and after.
SCORAD | At weeks 4 after the patient's admission
  The SCORAD score was calculated based on the types of lesions and body areas and was assessed separately for the head, neck, arms, legs, anterior trunk, back, and genitalia based on the area of skin involved and the severity of erythema, exudation, crusting, lichenification, and dryness. The scores report the severity of the patients' symptoms, with a total score ranging from 0 to 103, scores of 25 or lower indicating mild severity, scores of 26 to 50 indicating moderate severity, and scores of 51 to 103 indicating severe severity.. Patients were monitored for changes in SCROAD during treatment, observed for improvement in atopic dermatitis, and changes in points were calculated and compared before and after.

SECONDARY OUTCOMES:
Clinical Dermatologist Evaluation Form | At weeks 0, 2 and 4 after the patient's admission
  At weeks 0, 2 and 4 after the patient's admission, the clinician assessed the skin condition of the patient's entire face on a scale of 0-4 for each of the four indicators: erythema, erythema, papules, edema and desquamation.
Patient Self-Assessment Questionnaire | At weeks 0, 2 and 4 after the patient's admission
  Patients were asked to fill in the skin sensory self-assessment questionnaire at week 0, week 2 and week 4 after admission to the group to understand the improvement of their subjective symptoms.
Drug-Related Adverse Events. | through study completion, an average of 1.5years
  The onset, duration, severity, management, and consequences of adverse events related to the study drug were recorded and their relationship to the use of the study drug was determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Wang P, Wei X, Cheng L, Guo D, Du T, Guo W, Xi R, Duan Y, Liu X, Wang Y, Lu H, Yan G, Zhu J, Hua L, Li F. Efficacy and safety of BSZY cream for mild-to-moderate atopic facial dermatitis: protocol of a randomised, double-blind, controlled trial. BMJ Open. 2025 Mar 22;15(3):e087149. doi: 10.1136/bmjopen-2024-087149. PMID 40122554